CLINICAL TRIAL: NCT04305236
Title: A Phase II Open Label Trial of Neo-Adjuvant Abemaciclib With Fulvestrant in Patients Who Develop Localized Recurrence While on Adjuvant Endocrine Therapy With Molecular Evidence of Endocrine Resistance
Brief Title: Neo-Adjuvant Abemaciclib With Fulvestrant in Patients With ER/PR +HER Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted due to study funding
Sponsor: University of California, Irvine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Ritesh Parajuli, Assistant Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 18-79 [HS# 2020-5660]; 2020-5660 (Other: University of California, Irvine)
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Breast Neoplasm; Hormone Receptor Positive Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib and Fulvestrant (Experimental): Abemaciclib will be administered orally at the dose of 150 mg twice daily. Fulvestrant will be administered intramuscularly at an initial loading dose of 500mg on days 1 and 15 of the first cycle and then 500 mg intramuscularly every first day of each subsequent cycle. One cycle is 28 days.
  Interventions: Drug: Abemaciclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: VERZENIO™
Drug: Fulvestrant — Given Intramuscularly
  Other Names: FASLODEX®

SUMMARY:
This is a phase 2 single-arm, open-label determining efficacy of Neo-adjuvant Abemaciclib and Fulvestrant in subjects with Hormone receptor positive patients with localized non-metastatic breast cancer who develop local recurrence while on adjuvant endocrine therapy with molecular evidence of endocrine resistance.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of HR+ breast cancer. To fulfill the requirement of HR+ disease, a breast cancer must express, by immunohistochemistry (IHC), at least one of the hormone receptors (ER, progesterone receptor [PgR]) as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines (Hammond et al. 2010):

  1. For ER and PgR assays to be considered positive, ≥1% of tumor cell nuclei must be immunoreactive by immunohistochemistry (IHC) (Hammond et al. 2010).
* Patients must have Loco regional breast cancer (Stage I, Stage II and stage III per AJCC 8th edition criteria for staging of breast cancer)
* Patients must have localized recurrence while on adjuvant endocrine therapy
* Patients must have any known molecular evidence of endocrine resistance by next generation sequencing
* Age ≥ 18 years.
* ECOG performance status 0-1
* Have post-menopausal status as defined by following:

  1. Prior bilateral oophorectomy
  2. Age ≥ 60 years
  3. Age < 60 and amenorrheic (non-treatment-induced amenorrhea secondary to tamoxifen, toremifene, ovarian suppression, or chemotherapy) for at least 12 months. Follicle-stimulating hormone (FSH) and estradiol must be in the postmenopausal range.
* Have at least one measurable disease as defined per RECIST 1.1
* Adequate organ and marrow function as defined below:

  1. Hemoglobin* > 8 g/dL
  2. Absolute neutrophil count ≥ 1,500/mcL
  3. Total bilirubin ≤ 1.5 X institutional ULN, Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted
  4. AST (SGOT)/ALT (SPGT) ≤ 2.5 X institutional ULN
  5. Creatinine ≤ 1.5 X institutional ULN

     1. *Patients may receive transfusion of packed red blood cells (PRBC) to achieve this hemoglobin level at the discretion of the investigator; however, initial study drug treatment must not begin earlier than the day after the PRBC transfusion.
* Able to swallow oral medications
* Patients who received adjuvant radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and screening for the study.
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to enrollment. A washout period of at least 21 days is required between last chemotherapy dose and enrollment (provided the patient did not receive radiotherapy).
* Any known markers of response or resistance to CDK 4/6 inhibitors to be present in the biopsy specimen
* If patients have been treated with prior Neo-Adjuvant chemotherapy at the time of primary diagnosis and not at the time of recurrence, they will be included in the study.
* Must be able to sign a written informed consent, are reliable, willing to be available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Stage IV metastatic breast cancer

  1. This study will utilize the American Joint Committee on Cancer (AJCC) staging system, eight edition that provides a strategy for grouping patients with respect to prognosis. The AJCC has designated staging by TNM classification. The researchers will also review tumor size, lymph node status, and estrogen-receptor and progesterone-receptor levels in the tumor tissue.
* Patients with HER2 positive and triple negative breast cancer

  1. To fulfill the requirement of HER2- and Triple negative disease, a breast cancer must not demonstrate, at initial diagnosis or upon subsequent biopsy, overexpression of HER2 or should not express ER or PR receptors by either IHC or in-situ hybridization (ISH) as defined in the relevant ASCO/CAP guidelines (Wolff et al. 2013).
* Inflammatory breast cancer
* Newly diagnosed endocrine naïve patients
* No molecular evidence of endocrine resistance
* Prior treatment with any CDK 4/6 inhibitor and/or Fulvestrant
* Pre-menopausal women
* Are currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged not to be scientifically or medically compatible with this study. If a patient is currently enrolled in a clinical trial involving non-approved use of a device, then agreement with the principal investigator is required to establish eligibility
* Have had major surgery within 14 days prior to enrollment to allow for post-operative healing of the surgical wound
* Have initiated bisphosphonates or approved RANK ligand therapy for breast cancer with osseous metastasis, if patients are received Zolendronic acid or Denosumab in the adjuvant manner then such patients will be allowed participate
* Have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study (for example, history of major surgical resection involving the stomach or small bowel or preexisting Crohn's disease or ulcerative colitis , interstitial lung disease, severe dyspnea at rest, any pre-existing chronic condition resulting in baseline grade 2 or higher diarrhea)
* Have a personal history of any of the following conditions: syncope or cardiovascular etiology, ventricular tachycardia, ventricular fibrillation or sudden cardiac arrest
* Have a history of any other cancer (except for non-melanoma skin cancer or carcinoma in situ of the cervix) unless in complete remission with no therapy for a minimum of three years or have received an autologous or allogeneic stem-cell transplant
* Have an active bacterial or fungal infection or a detectable viral infection (for example HIV or viral hepatitis). Screening is not required for enrollment
* Recent therapy with a biologic agent or a monoclonal therapy is excluded. Wash out of at least three half-lives of monoclonal antibody would be required to be enrolled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Parajuli, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abemaciclib and Fulvestrant
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Abemaciclib and Fulvestrant
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Pathological Complete Response
Description: This is defined as the percentage of subjects who achieve a pathological complete response (pCR). A pCR is defined by no evidence of tumor cells in the final surgical specimen.
Time Frame: From start of study treatment to surgery, on average we expect 6 months.
Population: Data not collected
Arm/Group | Abemaciclib and Fulvestrant
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Response Rate
Description: To assess the overall response rate to the combination of Abemaciclib and Fulvestrant. Overall response rate (ORR) is defined as confirmed complete response (CR) and partial response (PR). Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1): Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. ORR = CR + PR
Time Frame: From start of study treatment to surgery, on average we expect 6 months.
Population: Data not collected
Arm/Group | Abemaciclib and Fulvestrant
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants Who Undergo Breast Conserving Surgery
Description: This is defined as the percentage of subjects who undergo breast conserving surgery after receiving Abemaciclib and Fulvestrant
Time Frame: From start of study treatment to surgery, on average we expect 6 months.
Population: Percentage of participants could not be analyzed due to early study termination.
Arm/Group | Abemaciclib and Fulvestrant
Number analyzed (Participants) | 0

4. Secondary Outcome: Recurrence Disease Free Survival
Description: Recurrence disease free survival will be defined as the time from surgery until patient develops recurrence.
Time Frame: Up to 5 years
Population: Data not collected
Arm/Group | Abemaciclib and Fulvestrant
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Grade 3-5 Adverse Events
Description: To evaluate the safety and tolerability of administering Abemaciclib and Fulvestrant. Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.
Time Frame: From start of study treatment to surgery, on average we expect 6 months.
Population: Refer to the adverse event table for specifics. There were no reported adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Abemaciclib and Fulvestrant
Number analyzed (Participants) | 1
percentage of participants | 0

6. Secondary Outcome: Percentage Change in Ki 67
Description: Percentage change in the Ki 67 will be evaluated from baseline to the treated specimen after breast surgery
Time Frame: From start of study treatment to surgery, on average we expect 6 months.
Population: Data not collected.
Arm/Group | Abemaciclib and Fulvestrant
Number analyzed (Participants) | 0

7. Secondary Outcome: Preoperative Endocrine Prognostic Index Score
Description: The preoperative endocrine prognostic index (PEPI) Score is a score that is used in clinical trials to assess response to Neo-Adjuvant endocrine therapy. The PEPI score takes into account the tumor and nodal stage, level of ER expression and Ki 67 following neoadjuvant endocrine therapy.
Time Frame: From start of study treatment to surgery, on average we expect 6 months.
Population: Data not collected.
Arm/Group | Abemaciclib and Fulvestrant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment to surgery, on average we expect 6 months.
Description: Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.
Arm/Group | Abemaciclib and Fulvestrant
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early study termination and depleted funding lead to the small number of patients enrolled onto the study. This also contributed to the inability to analyze the primary and secondary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT04305236/Prot_SAP_ICF_000.pdf